CLINICAL TRIAL: NCT07241767
Title: An Open Label, Multicenter Phase II Clinical Study on the Safety, Tolerability, and Efficacy of FH-006 Injection Combined With Other Anti-tumor Therapies in Lung Cancer Subjects
Brief Title: A Phase II Clinical Study of FH-006 for Injection Combined With Other Anticancer Therapies in Subjects With Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH-006-201-LC
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental)
  Interventions: Drug: FH-006 ; SHR-1316 ; BP102 ; Cisplatin ; Carboplatin
- Part B (Experimental)
  Interventions: Drug: FH-006 ; SHR-1316 ; BP102

INTERVENTIONS:
Drug: FH-006 ; SHR-1316 ; BP102 ; Cisplatin ; Carboplatin — FH-006 ; SHR-1316 ; BP102 ; Cisplatin ; Carboplatin
  Arms: Part A
Drug: FH-006 ; SHR-1316 ; BP102 — FH-006 ; SHR-1316 ; BP102
  Arms: Part B

SUMMARY:
Evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of FH-006 in combination with other anti-tumor treatments in lung cancer subjects, and determine the recommended dose (RP2D) and initial efficacy for phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years old (including both ends), gender is not limited.
2. Subjects with locally advanced or metastatic non-small cell lung cancer confirmed by histology or cytology as unsuitable for radical surgery or radiotherapy treatment
3. ECOG score is 0 or 1
4. Expected survival period ≥ 12 weeks
5. According to the RECIST v1.1 standard, there must be at least one measurable lesion.
6. Good level of organ function
7. The patient voluntarily joined this study and signed informed consent
8. Left ventricular ejection fraction (LVEF) ≥ 50%

Exclusion Criteria:

1. Suffering from other malignant tumors within the past 5 years
2. Subjects with active central nervous system (CNS) tumor metastasis, a history of meningeal metastasis, or current meningeal metastasis
3. Patients with uncontrollable tumor related pain
4. Has serious cardiovascular and cerebrovascular diseases
5. Significant clinically significant bleeding symptoms occurred within 3 months prior to the first study medication
6. Uncontrollable third interstitial fluid accumulation within 2 weeks of initial study medication
7. History of clinically significant pulmonary diseases
8. Receive other anti-tumor treatments within 4 weeks before the first medication
9. Severe infection within 4 weeks before the first medication
10. Active, known or suspected autoimmune diseases, and a history of autoimmune diseases.
11. History of immunodeficiency
12. Individuals with active pulmonary tuberculosis infection within the year prior to enrollment
13. Chest radiation therapy patients who received>30 Gy within 24 weeks prior to the first use of the investigational drug
14. The adverse reactions of previous anti-tumor treatments have not yet recovered to ≤ Grade I
15. Surgical treatment of important organs within 4 weeks prior to the first use of medication
16. Use attenuated live vaccine within 28 days prior to the first use of the investigational drug
17. There are other serious physical or mental illnesses or laboratory abnormalities present
18. Pregnant, lactating women, or female participants who plan to become pregnant within 14 months after the last use of the investigational drug during the study period
19. Having bleeding tendency, high risk of bleeding, coagulation dysfunction or thrombophilia tendency
20. Previously experienced hypertensive crisis or hypertensive encephalopathy
21. Suffering from significant vascular disease within 6 months prior to the first use of medication
22. Have undergone a biopsy or other minor surgery within 7 days prior to the first use of medication
23. Having severe, unhealed wounds, active ulcers, or untreated fractures
24. Gastrointestinal perforation occurred within 6 months prior to the first use of medication
25. 24-hour proteinuria quantification ≥ 1g within 7 days before the first medication
26. CT/MRI indicates tumor surrounding or invading large blood vessels

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
DLT (Dose-limiting toxicity)：Severe toxicity occurred 21 or 28 days after each subject received their first systemic anticancer treatment. | 21or28 days after the first administration of each subject
Incidence of Treatment-Emergent Adverse Events | from first dose to disease progression or death, up to 3 years.
RP2D (Recommended Phase II Dose)：This was determined through a comprehensive evaluation of safety data and pharmacokinetic characteristics. | from first dose to disease progression or death, up to 3 years
  This was determined through a comprehensive evaluation of safety data and pharmacokinetic characteristics.
ORR (Objective Response Rate) | from first dose to disease progression or death, whichever comes first, up to 3 years
  The proportion of patients whose tumor volume shrank to the pre-defined standard (complete or partial response) after treatment.

SECONDARY OUTCOMES:
Duration of response (DoR) | from first dose to disease progression or death, whichever comes first, up to 3 years
disease control rate (DCR) | from first dose to disease progression or death, whichever comes first, up to 3 years
progression free survival (PFS) | from first dose to disease progression or death, whichever comes first, up to 3 years
overall survival (OS) | from first dose to disease progression or death, whichever comes first, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided